CLINICAL TRIAL: NCT04554667
Title: Feasibility and Safety of Heavy Lifting Strength Training in Head and Neck Cancer Survivors Post-Surgical Neck Dissection
Brief Title: Heavy Lifting Strength Training in Head and Neck Cancer Survivors
Acronym: LIFTING
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-0169
Record Dates: First submitted 2020-09-11; First posted 2020-09-18 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Cancer of Head and Neck
Keywords: surgery; neck dissection; strength training; survivors; exercise
MeSH Terms: conditions — Head and Neck Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single arm, safety and feasibility trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Intervention (Experimental): Single exercise arm
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — Heavy Lifting Strength Training

SUMMARY:
The LIFTING trial will examine the feasibility and safety of a heavy lifting strength training (HLST) program in head and neck cancer survivors (HNCS) at least 1 years post surgical neck dissection. The trial will determine whether this training style is safe and feasible in HNCS. Physical and psychosocial changes will also be reported.

DETAILED DESCRIPTION:
RATIONALE Despite improvements in treatments, HNCS still endure numerous acute and chronic side effects. Strength training has been shown to manage some of these side effects but most interventions have involved light-to-moderate resistance training programs. HLST may produce better outcomes but it is unknown if such a weight training program is feasible and safe for HNCS.

OBJECTIVE The primary aim of this proposed study is to examine the feasibility and safety of a HLST program in HNCS at least 1 year post-surgical neck dissection.

METHODS This single arm feasibility study will recruit 15-20 HNCS to complete the HLST program 2 times per week. The primary feasibility outcomes will include the eligibility rate (with reasons for ineligibility), recruitment rate (with reasons for refusal), 1 repetition maximum testing rate (with reasons for not completing the test), program adherence (including attendance, dose modifications, and progression), and follow-up assessment rate (with reasons for drop out). The primary efficacy outcome will be strength gains from baseline. Secondary efficacy outcomes will include physical functioning, quality of life, fear of cancer recurrence, pain, body composition, anxiety, fatigue, stress, shoulder mobility, self-esteem, sleep, and motivation to engage in a HLST program.

SIGNIFICANCE Weight training is an effective intervention in HNCS but the optimal weight training prescription is unknown. If heavy weight training is deemed safe and feasible in HNCS, it can be compared to light-to-moderate load weight training to determine if it is a better prescription for improving outcomes that are important to HNCS.

ELIGIBILITY:
Inclusion Criteria:

* previously diagnosed with any subtype and stage of head and neck cancer
* at least one year post surgical neck dissection for head and neck cancer and showing full shoulder range of motion or recovery of the spinal accessory nerve
* adults ages 18 and older
* no unmanaged medical conditions, alcohol, and drug abuse
* approved for a heavy lifting strength training program by the treating surgeon and a certified exercise physiologist
* ability to understand and communicate in English

Exclusion Criteria:

* having comorbidities or uncontrolled medical conditions that their referred clinicians indicate as inappropriate to participate in exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Over 12 weeks
  Recruitment rate (with reasons for refusal).
  Recruitment minimum: 15 participants Recruitment maximum: 20 participants Higher number= better and more data
Muscular Strength | Changes from baseline to 12 weeks
  Change in muscular strength from baseline to postintervention with be assessed using maximal strength tests.
  Minimum: none Maximum: none Higher score= better strength
Program Adherence | Over 12 weeks
  Program adherence minimum: 80% Program adherence maximum: 100% Higher score= better adherence

SECONDARY OUTCOMES:
Physical functioning | Changes from baseline to 12 weeks
  Assessed using the Neck Dissection Impairment Index (NDII) and maximum strength tests.
  Minimum: 40 Maximum: 100 Higher score= worse impairment
Fear of cancer recurrence | Changes from baseline to 12 weeks
  Assessed using the Fear of Cancer Recurrence Inventory (FCRI)
  Minimum: 0 Maximum: 36 Higher score= worse fear of cancer recurrence
Post Traumatic Growth after cancer | Changes from baseline to 12 weeks
  How cancer has changed an individual's life will be assessed using the Post Traumatic Growth Inventory (PTGI)
  Minimum: 0 Maximum: 105 Higher score= better (positive) post traumatic growth transformation
Waist to hip ratio (body composition) | Changes from baseline to 12 weeks
  Assessed using waist to hip ratio (WHR) measure.
  Minimum WHR: none Maximum WHR: none Higher score WHR= worse body composition
Anxiety | Changes from baseline to 12 weeks
  Assessed using the Spielberger State Trait Anxiety Inventory (STAI)
  Minimum: 20 Maximum: 80 Higher score= worse anxiety
Fatigue | Changes from baseline to 12 weeks
  Assessed using the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) questionnaire
  Minimum: 0 Maximum: 52 Higher score=worse fatigue
Stress | Changes from baseline to 12 weeks
  Assessed using the Perceived Stress Scale (PSS)
  Minimum: 0 Maximum: 56 Higher score=worse perceived stress
Shoulder Mobility | Changes from baseline to 12 weeks
  Changes in shoulder mobility
  Minimum: 150 degrees (18-50 years); 130 degrees (over 50 years) Maximum: none Higher score= better mobility
Self-Esteem | Changes from baseline to 12 weeks
  Changes in level of self-esteem assessed using Rosenberg Self-Esteem (RSE) scale
  Minimum: 10 Maximum: 40 Higher score= better self-esteem
Sleep | Changes from baseline to 12 weeks
  Changes in sleep patterns assessed using the insomnia severity index (ISI)
  Minimum: 0 Maximum: 28 Higher score= worse insomnia
Motivation | Changes from baseline to 12 weeks
  Questions based on the theory of planned behaviour
  Minimum: 7 Maximum: 35 Higher score= better motivation
Cancer specific quality of life | Changes from baseline to 12 weeks
  Assessed using the Functional Assessment of Cancer Therapy-Head and Neck (FACT-H&N Symptom Index)
  Minimum: 0 Maximum: 40 Higher score= worse head and neck cancer symptoms
Cancer Symptom Burden | Changes from baseline to 12 weeks
  Assessed using the revised Edmonton Symptom Assessment System (ESAS-r)
  Minimum: 0 Maximum: 100 Higher score= worse cancer symptoms
Height | Changes from baseline to 12 weeks
  Assessed using standing height without shoes.
  Minimum height: none Maximum height: none Taller: not specifically better or worse
Weight | Changes from baseline to 12 weeks
  Assessed using a digital scale without shoes.
  Minimum weight: none Maximum weight: none Higher weight: typically worse, but depends on other factors (ie. height, muscle mass, overall health status)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S Courneya, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ntoukas SM, McNeely ML, Seikaly H, O'Connell D, Courneya KS. Feasibility and safety of Heavy Lifting Strength Training in Head and Neck Cancer survivors post-surgical neck dissection (the LIFTING trial). Support Care Cancer. 2023 May 22;31(6):348. doi: 10.1007/s00520-023-07815-2. PMID 37212970